CLINICAL TRIAL: NCT01476332
Title: A Single Dose (Part 1) and Multiple Dose (Part 2) Phase I, Double-blind, Placebo-controlled, Safety, Tolerability and Pharmacokinetic Study of 0.5% and 2.5% Cis-UCA Eye Drops in Adult Healthy Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of 0.5% and 2.5% Cis-UCA Eye Drops in Adult Healthy Volunteers (Phase I)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laurantis Pharma, Ltd. (Industry)
Collaborators: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL11001; 2011-004283-30 (EudraCT Number)
Record Dates: First submitted 2011-11-10; First posted 2011-11-22 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Dry Eye
Keywords: eyes; cis-urocanic acid; safety; tolerability; pharmacokinetics
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: Cis-UCA 0.5% eye drops (Experimental)
  Interventions: Drug: cis-urocanic acid 0,5% eye drops
- Group 2: Cis-UCA 2.5% eye drops (Experimental)
  Interventions: Drug: cis-urocanic acid 2.5% eye drops
- Group 3: Placebo for cis-UCA, eye drops (Placebo Comparator)
  Interventions: Drug: Placebo for cis-UCA, eye drops

INTERVENTIONS:
Drug: cis-urocanic acid 0,5% eye drops — one drop three times a day, applied on one eye at Part 1 and on both eyes at Part 2
  Arms: Group 1: Cis-UCA 0.5% eye drops
Drug: cis-urocanic acid 2.5% eye drops — one drop three times a day, applied on one eye at Part 1 and on both eyes at Part 2
  Arms: Group 2: Cis-UCA 2.5% eye drops
Drug: Placebo for cis-UCA, eye drops — one drop three times a day, applied on one eye at Part 1 and on both eyes at Part 2
  Arms: Group 3: Placebo for cis-UCA, eye drops

SUMMARY:
The purpose of this two-part study is to evaluate safety, tolerability and pharmacokinetics of 0.5% and 2.5% cis-UCA eye drops in comparison to placebo in adult healthy volunteers.

DETAILED DESCRIPTION:
This is a Phase I single-centre, double-blind, placebo-controlled, single and multiple dose study to evaluate safety, ocular tolerability and pharmacokinetics of 0.5% and 2.5% cis-UCA eye drops in healthy volunteers for up to 15 days. After the single day dose (three times) on day 1 and the subsequent 7 (± 1) days wash-out period, a multidose phase with three times a day administration for 14 days will start

Primary objectives:

* Part 1: To evaluate the safety and ocular tolerability of 0.5% and 2.5% cis-UCA eye drops and placebo for cis-UCA eye drops when administered on a randomized eye three times during a single day, assessed up to 7 (± 1) days following dosing in healthy volunteers
* Part 2: To evaluate the safety and ocular tolerability of 0.5% and 2.5% cis-UCA eye drops and placebo for cis-UCA eye drops when administered on both eyes three times a day for 14 days, assessed up to 7 days following the last dosing in healthy volunteers

Secondary objectives:

* To evaluate single dose pharmacokinetics of 0.5% and 2.5% cis-UCA eye drops when administered on a randomized eye in adult healthy volunteers
* To evaluate the pharmacokinetics of 0.5% and 2.5% cis-UCA eye drops when administered on both eyes three times a day for 14 days in adult healthy volunteers

Healthy male or female volunteer, 18-65 years of age, with no history of significant eye disease or any current eye disease that would affect the pharmacokinetics of cis-UCA. Subjects without any treatment-emergent adverse events during Part 1 may continue to Part 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained prior to any screening procedure
* Caucasian male or female subject
* Age 18-65 y
* Weight at least 45 kg
* Corrected visual acuity > 20/25 in both eyes
* Intraocular pressure < 21 mmHg, with a difference between eyes of < 4 mmHg
* Ability to tolerate and self-administer vehicle eye drops
* Normal slit lamp examination and dilated fundoscopic examination
* Normal clinical laboratory profiles, defined as complete blood count, serum chemistry, and urinalysis values within the normal range
* Willingness to abstain from concomitant use of ocular or systemic medication (excluding oral contraceptives, ibuprofen, paracetamol, calcium preparations and vitamins) from 2 weeks prior to the start of study dosing until study completion
* Willingness to comply with study-related procedures
* Negative urine pregnancy test (premenopausal female subject) at screening and use of adequate contraceptive measures throughout the study and 30 days after the last study medication dose
* A premenopausal female subject should be either surgically sterile or using a reliable contraception method: intrauterine device; oral combination pill or hormonal contraception patch; or two of the following: intra-vaginal hormonal ring, oral contraceptive containing progestin only, spermicidal foam, condom, sterilization of male sexual partner (surgical vasectomy)
* Subject with no current heterosexual relationship may be included according to the judgment of the Investigator
* If menopause occurred 2 years ago at the minimum, no contraception is required for a female participant, nor pregnancy test
* Reliable contraception for a male subject is concordant with above listed methods for females, as applicable

Exclusion Criteria:

* History of ocular surgery, trauma, or chronic ocular disease
* Current use of contact lenses or discontinuation of contact lens use within 2 weeks of the first dosing day
* Any ocular abnormalities or ocular symptoms (defined as a non-zero score on assessment scales)
* Use of ocular agents (including all types of eye drops) within the past month prior to the first dosing day or anticipated use of ocular agents during the study period
* Use of systemic or inhaled nasal or pulmonary corticosteroids within the past month prior to the first dosing day
* Use of systemic antihistamines within one week prior to the first dosing day
* History or evidence of ocular infection, inflammation, blepharitis, or conjunctivitis within 2 months prior to the first dosing day; history of herpes simplex keratitis at any time
* Current ocular allergy symptoms
* Loss, donation, or removal of 400 ml or more of blood within 2 months prior to the first dosing day
* Women who are pregnant or breastfeeding, or non-sterile or premenopausal women who refuse to use two proven methods of contraception during the study and for at least 30 days following the final dose of study drug
* Participation in another clinical drug or device study within 2 months prior to the first dosing day
* Current smoking
* Current or history of drug or alcohol abuse
* Known human immunodeficiency virus- or acquired immunodeficiency syndrome -related illness.
* Allergy to cis-UCA, or any constituents of the cis-UCA eye drops (cis-urocanic acid, aqua, sodium chloride, polyvinyl alcohol, sodium hydroxide, and/or hydrochloric acid) or placebo for cis-UCA eye drops (aqua, sodium chloride, polyvinyl alcohol, sodium hydroxide, and/or hydrochloric acid)
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, would affect the subject's ability to follow study-related procedures, or may interfere with the interpretation of study results and, in the Investigator's opinion, would make the subject inappropriate for entry into this study.
* Doubtful availability to complete the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
IER (Institute of Eye Research) grading scale evaluates bulbar conjunctival redness, lid redness and corneal staining and extent | 36 days

SECONDARY OUTCOMES:
Ocular comfort rating | 36 days
Early Treatment Diabetic Retinopathy Study table, a visual acuity test | 36 days
Anterior chamber cells and flare using SUN Working Group Grading Schemes | 36 days
Ocular pressure | 36 days
Schirmer's test | 36 days

CONTACTS AND LOCATIONS:
Overall Officials: Kai Kaarniranta, Professor, Principal Investigator — Kuopio University Hospital, Department of Ophthalmology
Locations (1):
- Kuopio University Hospital, Department of Ophthalmology, Kuopio, Finland